CLINICAL TRIAL: NCT06598059
Title: A Pivotal, Prospective, Multicentre, Single-arm Study Evaluating the Safety and Efficacy of a Dexamethasone Eluting Slim Modiolar Electrode Array (EA32D).
Brief Title: Safety and Efficacy of a Drug Eluting Slim Modiolar Electrode Array
Acronym: DEE-REX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: University of Iowa (Other); LWB Consulting (Unknown); Althea Anagnostopoulos Harrington (Unknown); MV Clinical Research, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5849
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss
Keywords: cochlear implant; dexamethasone; fibrosis
MeSH Terms: conditions — Hearing Loss; Fibrosis | interventions — Cochlear Implants; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Drug-eluting electrode array (CI632D) (Experimental): Participants will be implanted with the slim modiolar dexamethasone-eluting electrode array.
  Interventions: Device: Cochlear implant; Drug: Dexamethasone

INTERVENTIONS:
Device: Cochlear implant — CI632D cochlear implant
  Other Names: CI632D; Slim modiolar dexamethasone-eluting electrode array
Drug: Dexamethasone — CI632D, dexamethasone-eluting cochlear implant
  Other Names: CI632D; Slim modiolar dexamethasone-eluting electrode array

SUMMARY:
This clinical study will test a new type of cochlear implant known as CI632D. This experimental cochlear implant has been designed to slowly release a drug called dexamethasone. Dexamethasone works to ease inflammation and reduce tissue injury, which is common after any type of surgery. The goal is to learn if the dexamethasone in the CI632D implant lessens these reactions inside the ear following surgery and if this makes the implant work as well, or even better, in improving hearing than what would be expected with a standard cochlear implant. The study will be conducted in adults with sensorineural hearing loss, a type of hearing loss caused by damage to the inner ear or auditory nerve (the nerve that carries sound signals from the ear to the brain). The study participants will receive the CI632D experimental implant and will complete tests to see how well they are hearing and how well the implant is working.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, at time of consent.
* Postlinguistic moderately severe to profound sensorineural hearing loss, defined by a four frequency (500, 1000, 2000, 4000 Hz) pure-tone average unaided threshold (PTA4) ≥ 60 decibels hearing level (dB HL), in the ear to be implanted (For this study, moderately severe is defined by a four-frequency, pure-tone average threshold (PTA4) over the range 500 through 4000 Hz of more than 55 dB HL through 70 dB HL, inclusive. Profound is defined by a PTA4 of more than 90 dB HL).
* Pure-tone average unaided threshold (500 through 4000 Hz) ≥ 30 dB HL, in the contralateral ear.
* Preoperative aided word score ≤ 40% correct in the ear to be implanted.
* Evidence of pneumococcal vaccination (e.g., Pneumovax) according to local guidelines.
* Candidate is proficient in the language used to assess speech perception performance.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Intra-axial (within the brain) lesions or deafness due to lesions of the acoustic nerve affecting the ear to be implanted.
* Middle ear infection (including acute otitis media, chronic otitis media, suppurative otitis media, or serous drainage) in the ear to be implanted either at the time of surgery or within 3 months prior to enrolment.
* Active autoimmune disease or active immunosuppressive therapy.
* Presence of a tympanic membrane perforation or a history of otologic surgery within 3 months prior to enrolment, in the ear to be implanted.
* Previously reported diagnosis of auditory neuropathy, in the ear to be implanted.
* Previously reported diagnosis, in the ear to be implanted, of Large Vestibular Aqueduct Syndrome (LVAS), Meniere's disease, or cochlear hydrops.
* Ossification, otosclerosis, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, in the ear to be implanted.
* Current cerebrospinal fluid (CSF) shunts or drains, existing perilymph fistula, skull fracture or CSF leaks.
* Previously reported diagnosis of bacterial meningitis.
* Known allergic reaction or contraindication to dexamethasone or corticosteroids.
* Severe, or poorer, bilateral sensorineural hearing loss prior to 5 years of age, as reported by the subject. (For this study, severe is defined by a PTA4 of more than 70 dB HL through 90 dB HL, inclusive).
* Severe, or poorer, sensorineural hearing loss for more than 20 years, as reported by the subject, in the ear to be implanted.
* Prior cochlear implantation in either ear.
* Medical plan for cochlear implantation during the clinical investigation, contralateral to the ear to be implanted.
* Medical or psychological conditions that contraindicate general anaesthesia, surgery, or participation in the clinical investigation as determined by the Investigator.
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations inherent to the surgical procedure(s) and prosthetic devices, as determined by the Investigator.
* Women who are pregnant.
* Additional disabilities that may affect the subject's participation or safety during the clinical investigation.
* Unable or unwilling to comply with all the requirements of the clinical investigation as determined by the investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device unless Cochlear sponsored and determined by Investigator or Sponsor to not impact this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Coprimary endpoint 1: Mean monopolar 1 plus 2 (MP1+2) impedances (kOhms) at 3 months postactivation | On day of implantation and at 1- and 3-months postactivation
  Impedance will be measured across the active electrodes of the implant for each participant.
Coprimary endpoint 2: Mean change in word recognition score in the best unilateral listening mode in quiet from preimplantation to 3 months postactivation | Preoperative baseline and 3-months postactivation
  Within-subject change in consonant-nucleus-consonant (CNC) words in quiet (% correct) calculated as the average across 2 runs of the test conducted on each participant. CNC word score ranges from 0-100%, higher the score the better the outcome.

SECONDARY OUTCOMES:
Mean within-subject change in the global score of the Speech, Spatial, and Qualities of hearing scale (SSQ12) from preimplantation to postimplantation | Preoperative baseline and 6-months postactivation
  Within-subject change in Global SSQ12 scores at 6-months postactivation compared with preoperative baseline. The global SSQ12 score ranges from 0-10, higher the score the better the outcome.
Mean within-subject change in sentence recognition score in the best unilateral listening mode in noise from preimplantation to postimplantation | Preoperative baseline and 6-months postactivation
  Within-subject change in AzBio sentence in noise score at a +10 dB Signal-to-Noise Ratio (SNR) at 6-months postactivation compared with preoperative baseline. AzBio score ranges from 0-100%, higher the score the better the outcome.
Mean within-subject change in sentence recognition score in the best bilateral listening mode in noise from preimplantation to postimplantation | Preoperative baseline and 6-months postactivation
  Within-subject change in AzBio sentence in noise score at a +10 dB Signal-to-Noise Ratio (SNR) at 6-months postactivation compared with preoperative baseline. AzBio score ranges from 0-100%, higher the score the better the outcome.

OTHER OUTCOMES:
Proportion of participants who experience an adverse event and the proportion of participants who experience a device deficiency throughout the study | From implantation to 12-months postimplantation (study end)
  Adverse events will be recorded as overall, by severity, by relatedness to device or procedure, or by seriousness. Device deficiency will be recorded as overall and by type.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Parkinson, PhD, Study Director — Cochlear
Locations (11):
- United States (11):
  - UCLA Medical Center, Los Angeles, California
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Iowa, Iowa City, Iowa
  - Henry Ford Health, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - NYU Langone Health, New York, New York
  - Northwell Health Long Island Jewish Medical Center, New York, New York
  - University Hospitals, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No